CLINICAL TRIAL: NCT06290323
Title: Effects of Postoperative Quadratus Lumborum Block on Sub-Urine System Symptoms in Ureteroscopic Lithotripsy Operations: Randomized Controlled Study
Brief Title: Effects of Quadratus Lumborum Block on Lower Urinary System Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Eylem Yaşar, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11/05/2022-9/VIII
Record Dates: First submitted 2024-02-12; First posted 2024-03-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lithotripsy; Lower Urinary Tract Symptoms; Pain
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Pain

STUDY DESIGN:
Intervention Model Description: Patients with double J catheter inserted into ureteroscopic lithotripsy surgeries due to urethral stones
Who Masked: Outcomes Assessor
Masking Description: The researcher evaluating the survey does not know which group the patients are.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Other): Patients in the first group are the control group, and after spinal anesthesia, the sensory block is formed, and the lithotomy position will be taken for the surgical procedure. Patients will be monitored for 48 hours for postoperative pain (Numarating Raiting Scala: NRS) and side effects. On the postoperative 7th day, the patient's pain level will be NRS, and the DJS-connected sub-urinary system symptoms assessed will be evaluated with the ureteral stent discomfort questionnaire (with the stent inserted). In our clinic, approximately one month after URS operations, control cystoscopy is performed and ureteral stents are removed. After five days of removal of the ureteral stent, the lower urinary system symptoms will be questioned with the ureteral stent discomfort questionnaire (after removal of the stent).
  Interventions: Procedure: Placebo
- Quadratus lumborum (Active Comparator): After the posterior quadratus lumborum block was made in the lateral decubitus position, the patient was taken to the lithotomy position for surgery. Patients will be monitored for 48 hours for postoperative pain (Numarating Raiting Scala: NRS) and side effects. On the postoperative 7th day, the patient's pain level will be NRS and the DJS-connected sub-urinary system symptoms will be assessed and evaluated using the ureteral stent discomfort questionnaire (with the stent inserted). In our clinic, approximately one month after URS operations, a control cystoscopy is performed, and ureteral stents are removed. After five days of removal of the ureteral stent, the lower urinary system symptoms will be questioned with the ureteral stent discomfort questionnaire (after removal of the stent).
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Quadratus lumborum block — Posterior quadratus lumborum block
  Arms: Quadratus lumborum
Procedure: Placebo — Patients in the first group are the control group and after spinal anesthesia, the sensory block is formed, the lithotomy position will be taken for the surgical procedure.
  Arms: Placebo

SUMMARY:
The most common reason for applying to a hospital in the postoperative period is due to the double J stent inserted during operations of the ureteroscopic lithotripsy, which is reflected pain (T11-L2). The posterior approximation QL block (QL-P) extends more quickly to the thoracic paravertebral cavity or thoracolumbar plane, creating analgesia from T 7' to L 1'. The effects of double J catheter in patients are followed by the 'Ureteral Stent Symptom Scoring Survey.' QL-P for postoperative analgesia after URS operations Our primary hypothesis in this prospective, randomized, controlled study is that the symptoms of the sub-urinary system associated with the DJS of the QL-P block will decrease. Our secondary hypotheses in the study are to investigate the effects of the unilateral QL-P block, made under ultrasound guidance, on pain scores after ureteroscopic lithotripsy operations due to unilateral ureteral stones made under spinal anesthesia.

DETAILED DESCRIPTION:
All patients will be seated to apply spinal anesthetic. Patients will be inserted into the interspinal space using a 25-gauge Quincke needle from the lumbar (L) 3-L4 spinal interval or the L4-L5 spinal interval, thereby inducing a sensory block at a 0.5% hyperbaric bupivacaine level with a Trocal (T) 10. Once a T-10 level sensory block has been established, the patients will be separated into two groups. As the control group, the individuals comprising Group 1 will be positioned in the lithotomy position after the sensory block for the surgical procedure. Group 2 patients will be placed in lateral decubitus to conduct a quadratus lumborum block. Once the skin's surface has been sterilized, the convex ultrasound probe (SonoSiteMTurbo; FUJIFILM SonoSite, Bothell, WA) will be moved laterally to the lateral to visualize the psoas and quadratus lumborum muscles. The probe will be inserted perpendicular to the spine in the 12th vertebral body. The in-plane method with the lateral of the probe 22 gauge needle, between the quadratus lumborum muscle and the front layer of the thoracolumbar fascia after the position accuracy is determined with 1-2 mL serum physiologic, %0.375 Mg of bupivacaine will be injected in 20 ml. The patient will then be placed in the lithotomy position for the surgical procedure. Patients of a blind research assistant to the group distribution are seen on-site in the 1st, 6th, 12th, and 24th hours after surgery, postoperative 7. Per phone daily, pain intensities will be assessed by a 'numerical assessment scale' (Numeric Rating Scala: NRS). If NRS is above 3 for half an hour, 100 mg tramadol will be added. For 48 hours, tramadol and non-steroidal anti-inflammatory consumption will be monitored. In addition, complications such as local anesthesia toxicity, allergy, internal organ injury, postoperative nausea and vomiting, and postoperative bleeding will be recorded. In addition, on the 7th post-operative day, the patient's pain level will be evaluated with NRS, and the sub-productive system symptoms connected to DJS are assessed with the ureteral stent symptom scoring questionnaire (while inserted in the stent). In our clinic, approximately one month after URS operations, a control cystoscopy is performed, and ureteral stents are removed. After five days of removal of the ureteral stent, the lower urinary system symptoms will be questioned with the ureteral stent symptom scoring questionnaire (after the stent is removed).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral URS planned to be applied
* DJS is planned to be inserted due to unilateral stone size of 5-15 mm.
* ASA I-II-III patients

Exclusion Criteria:

* Patients with bilateral ureteral stones,
* Patients with >15 mm or <5 mm ureteral stones,
* Patients with known paracetamol allergy,
* Patients with any contraindications to the regional technique
* Patients with chronic analgesic use
* Patients with a body mass index over 35 kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Quadratus posterior block | 1 month
  On the 7th post-operative day, lower urinary tract symptoms due to the ureteral stent will be evaluated with the ureteral stent symptom scoring questionnaire (with the stent in place) (questionnaire 1).
  Approximately one month after their operations, patients' lower urinary tract symptoms will be questioned withent symptom scoring survey (after stent removal) (survey 2) (Appendix 2) five the ureteral st days after their ureteral stents are removed.

SECONDARY OUTCOMES:
Pain Score | 7 days
  To evaluate the patients' postoperative pain scores (7 days) using the Numerical Rating Scale. If NRS is above 3 for half an hour, 100 mg tramadol will be added.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Yasar, MD, Principal Investigator — Mugla Sitki Kocman Training and Research Hospital
Locations (1):
- Mugla Sitki Kocman Training and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If any organization asks for our study data, we may share our data without revealing the identities of the patients.